CLINICAL TRIAL: NCT01784432
Title: Effects of Low-level Laser Therapy on Global Gene Expression of Young Males Submitted to Physical Strength Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Centro de Pequisas de Ótica e Fotônica (Other); Faculty of Medicine of Ribeirão Preto (FMRP-USP) (Other); Fundação Hemocentro de Ribeirão Preto (Unknown)
Responsible Party: Principal Investigator, Cleber Ferraresi, MSc, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 0150.0.135.000-10
Record Dates: First submitted 2012-09-15; First posted 2013-02-05 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: low-level laser therapy; muscle performance; strength training; gene expression; microarrays
MeSH Terms: interventions — Low-Level Light Therapy; Lasers; Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-level laser therapy and training (Active Comparator): Effects of low-level laser therapy on muscle performance during physical strength training and gene expression of muscle tissue.
  Interventions: Device: Low-level laser therapy and training
- Training without low-level laser therapy (Active Comparator): Effects of physical strength training without low-level laser therapy on muscle performance and gene expression of muscle tissue
  Interventions: Other: Training

INTERVENTIONS:
Device: Low-level laser therapy and training
  Other Names: Laser; Laser therapy; Low-level laser therapy
  Arms: Low-level laser therapy and training
Other: Training
  Arms: Training without low-level laser therapy

SUMMARY:
Muscle performance is largely influenced by modulations in gene expressions of muscle tissue. In this context, low-level laser therapy has been used to improve muscle performance in experimental models and human researches. Thereby, the investigators examined modulations on global gene expression of muscle tissue influenced by exercise associated to low-level laser therapy.

DETAILED DESCRIPTION:
This study assessed muscle performance in isokinetic dynamometry and leg press device; global gene expression of muscle tissue by microarray analysis

ELIGIBILITY:
Inclusion Criteria:

* healthy males aged between 18 and 28 years;
* body mass index (BMI) equal to or less than 26 kg/m2;
* moderated pattern of physical activity

Exclusion Criteria:

* previous injury to the femoral quadriceps or hamstring muscles (within 6 months prior to study),
* osseous or articular disorder in the lower limbs,
* cardiovascular system disorders,
* systemic disease, and
* taking prescription medicines or using dietary supplements such as muscle mass builders

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Global gene expression by microarray analysis | 12 weeks

SECONDARY OUTCOMES:
Muscle performance in leg press device | 12 weeks
Muscle performance in isokinetic dynamometer | 12 weeks

OTHER OUTCOMES:
Immunohistochemical analysis | 12 weeks
  Immunohistochemical analysis to quantify morphology and cells of muscle tissue as satellite cells.

CONTACTS AND LOCATIONS:
Overall Officials: Cleber Ferraresi, MSc, Principal Investigator — Universidade Federal de Sao Carlos; Nivaldo A Parizotto, PhD, Study Director — Universidade Federal de Sao Carlos; Vanderlei S Bagnato, PhD, Study Director — University of Sao Paulo
Locations (1):
- Federal University of São Carlos, São Carlos, São Paulo, Brazil

REFERENCES:
- [Background] Ferraresi C, de Brito Oliveira T, de Oliveira Zafalon L, de Menezes Reiff RB, Baldissera V, de Andrade Perez SE, Matheucci Junior E, Parizotto NA. Effects of low level laser therapy (808 nm) on physical strength training in humans. Lasers Med Sci. 2011 May;26(3):349-58. doi: 10.1007/s10103-010-0855-0. Epub 2010 Nov 18. PMID 21086010
- [Background] Vieira WH, Ferraresi C, Perez SE, Baldissera V, Parizotto NA. Effects of low-level laser therapy (808 nm) on isokinetic muscle performance of young women submitted to endurance training: a randomized controlled clinical trial. Lasers Med Sci. 2012 Mar;27(2):497-504. doi: 10.1007/s10103-011-0984-0. Epub 2011 Aug 26. PMID 21870127